CLINICAL TRIAL: NCT02095951
Title: Preemptive Ethanol Lock Therapy in Pediatric Hematology/Oncology Patients With Catheter Associated Bloodstream Infection: Impact on Length of Stay and Catheter Salvage
Brief Title: Preemptive Ethanol Lock Therapy in Pediatric Bloodstream Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Michigan (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Eric McGrath, Assistant Professor of Pediatrics - Clinical, Children's Hospital of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024.11
Record Dates: First submitted 2014-03-17; First posted 2014-03-26 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-08

CONDITIONS: Leukemia; Lymphoma; Blood Disorders; Solid Tumors
MeSH Terms: conditions — Leukemia; Lymphoma; Hematologic Diseases | interventions — Ethanol; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-emptive Ethanol Lock Therapy Group (Experimental): Participants receive ethanol lock before blood cultures grow germ
  Interventions: Drug: Ethanol lock therapy (ELT)
- Standard Ethanol Lock Therapy Group (Active Comparator): Participants receive ethanol lock if and only after blood cultures grow germ
  Interventions: Drug: Ethanol lock therapy (ELT)

INTERVENTIONS:
Drug: Ethanol lock therapy (ELT) — Participants will be randomized to receive early (preemptive) ELT (after 12 hours from time blood culture drawn, but before blood culture positive, R/O sepsis) with systemic antimicrobials versus standard ELT (placed in catheter when blood culture is positive for growth of a germ) with systemic antimicrobials.
  Other Names: 70% Ethanol in water

SUMMARY:
The study team will compare hospital length of stay (LOS) and attributable length of stay (ALOS, the LOS attributable to CRI), in a randomized, un-blinded prospective trial utilizing short-dwell ethanol-lock therapy (ELT) (4 hours to 24 hour dwell times per day, repeated for up to 72 hours) placed within 24 - 36 hours of admission(Group 1, Preemptive ELT) versus ELT placed at the time of first positive blood culture report (Group 2, Rescue ELT (Standard of Care ). ELT will be given in both groups, in combination with systemic antibiotics, for the treatment of CRI (suspected or proven) of the blood in children with central catheters. Participants will be enrolled from patients with hematologic/oncologic disorders and bone marrow or hematopoetic stem cell transplants (BMT) admitted for care to Children's Hospital of Michigan (CHM), a tertiary care pediatric hospital in Detroit, Michigan. ALOS will be defined as the number of hospital days between first symptoms of Catheter-related infection (CRI) (or date of admission for those admitted with symptoms) and first negative blood culture.

Study Hypothesis: The main hypothesis is that the short-dwell ethanol-lock therapy, defined above, placed within 24 - 36 hours of symptoms/admission (Arm 1) versus ELT placement at the time of first positive blood culture report (Arm 2), with concomitant systemic antibiotics, for the treatment of CRI (suspected or proven) of the blood in children with central catheters in the H/O/BMT population will have shorter hospital length of stay (LOS) and attributable LOS (ALOS) and therefore lower hospital costs.

DETAILED DESCRIPTION:
The study team will compare hospital length of stay (LOS) and attributable length of stay (ALOS, the LOS attributable to CRI), in a randomized, un-blinded prospective trial utilizing short-dwell ethanol-lock therapy (ELT) (4 hours to 24 hour dwell times per day, repeated for up to 72 hours) placed within 24 - 36 hours of admission(Group 1, Preemptive ELT) versus ELT placed at the time of first positive blood culture report (Group 2, Rescue ELT (Standard of Care ).

ELT will be given in both groups, in combination with systemic antibiotics, for the treatment of Catheter-related Infection (CRI) (suspected or proven) of the blood in children with central catheters. Participants will be enrolled from patients with hematologic/oncologic disorders and bone marrow or hematopoetic stem cell transplants admitted for care to Children's Hospital of Michigan (CHM), a tertiary care pediatric hospital in Detroit, Michigan. ALOS will be defined as the number of hospital days between first symptoms of CRI (or date of admission for those admitted with symptoms) and first negative blood culture.

Aim 1: Compare two different treatment regimens for CRI using ELT (the preemptive ELT vs. standard of care) by way of a prospective, randomized, two-arm study.

Study Hypothesis: The main hypothesis is that the short-dwell ethanol-lock therapy, defined above, placed within 24 - 36 hours of symptoms/admission (Arm 1) versus ELT placement at the time of first positive blood culture report (Arm 2), with concomitant systemic antibiotics, for the treatment of CRI (suspected or proven) of the blood in children with central catheters in the H/O/BMT population will have shorter hospital length of stay (LOS) and attributable LOS (ALOS) and therefore lower hospital costs.

Aim 2: Compare sterilization rate of the infected intravascular device after ethanol-lock therapy (as defined by a negative blood culture obtained from the infected catheter 24 - 72 hours after ELT) and central catheter salvage rate after CRI using ELT in the two study arms. If the central catheter is salvaged for further clinical use, recurrence of infection with the same organism (re-infection) of the central catheter for 28 days from date of first ELT procedure will also be assessed.

Aim 3: Assess tolerability and adverse effects of the ELT (safety).

Aim 4: Perform sub-group analysis on the BSI episodes meeting National Healthcare Safety Network (NHSN) criteria for laboratory confirmed central line associated BSI (CLABSI) into the three categories of Criteria 1, 2 or 3 within the pediatric

ELIGIBILITY:
Inclusion Criteria:

* All children up to 21 years of age, with central catheters (any type) that develop symptoms and are admitted to CHM with an underlying H/O/BMT diagnosis for individual episodes of suspected or proven CRI of the blood, including rule out sepsis, will be screened for potential participation in this study.
* Individual CRI episodes in the same patient will be defined as a distinct central catheter associated blood stream infection if separated by greater than 28 days from prior ELT procedure and caused by a different organism identified on culture than the prior central catheter associated blood stream infection episode.
* Participants meeting study enrollment criteria will be offered participation and must have parental full informed consent, adolescent assent and young child verbal assent prior to enrollment as applicable.

Exclusion Criteria:

* Children with documented allergy to ethanol or alcohol will be excluded. Blood cultures from patients that are reported positive for pathogen growth within 12 hours from the time they are obtained will be excluded from the study.
* Any patient at CHM with an infected central catheter and with another indwelling foreign body that communicates directly with the bloodstream, of which infection or colonization could not be excluded directly, will also be excluded from the study (i.e. Left Ventricular Assist Device) as it will not be possible to assess sterilization of the central catheter.
* Any patient with endocarditis or presumed endovascular infection will also be excluded.
* Any patient deemed critically ill or unstable, upon admission or during the early treatment course, in which case the treating clinician(s) feel that immediate line removal is potentially life-saving will be excluded from the study.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J McGrath, MD, Principal Investigator — Wayne State University
Locations (1):
- Children's Hospital of Michigan, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McGrath EJ, Salloum R, Chen X, Jiang Y, Boldt-MacDonald K, Becker C, Chu R, Ang JY. Short-dwell ethanol lock therapy in children is associated with increased clearance of central line-associated bloodstream infections. Clin Pediatr (Phila). 2011 Oct;50(10):943-51. doi: 10.1177/0009922811409568. Epub 2011 May 27. PMID 21622689
- [Background] Chaudhary M, Bilal MF, Du W, Chu R, Rajpurkar M, McGrath EJ. The impact of ethanol lock therapy on length of stay and catheter salvage in pediatric catheter-associated bloodstream infection. Clin Pediatr (Phila). 2014 Oct;53(11):1069-76. doi: 10.1177/0009922814533591. Epub 2014 May 7. PMID 24807976
- [Background] Rajpurkar M, McGrath E, Joyce J, Boldt-MacDonald K, Chitlur M, Lusher J. Therapeutic and prophylactic ethanol lock therapy in patients with bleeding disorders. Haemophilia. 2014 Jan;20(1):52-7. doi: 10.1111/hae.12241. Epub 2013 Aug 1. PMID 23906245
- [Result] McGrath E, Du W, Rajpurkar M. Preemptive Ethanol Lock Therapy in Pediatric Hematology/Oncology Patients With Catheter-Associated Bloodstream Infection: Impact on Length of Stay, Cost, and Catheter Salvage. Clin Pediatr (Phila). 2018 Mar;57(3):285-293. doi: 10.1177/0009922817717327. Epub 2017 Jun 30. PMID 28664750

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 135 episodes screened, but only 36 initially met enrollment criteria. 27 unique patients were enrolled for 33 episodes (6 patients enrolled twice) of possible catheter infection.
Pre-assignment Details: 3 enrolled participants were removed from the study/analysis for failure to meet final enrollment criteria. Patient participants could be re-enrolled in the study more than once if their infection episodes (cases) were separated by at least 28 days.
Units Other Than Participants: Catheter Infection Episodes (Cases)
Groups:
- Pre-emptive Ethanol Lock Therapy Group: Study intervention group (Arm 1). Received Early Ethanol Lock Therapy before blood culture results were reported as positive or negative.
- Standard Ethanol Lock Therapy Group: Standard of Care Group (Arm 2) that received Ethanol Lock Therapy if and only if the blood culture was positive for growth of an organism.
Period: Overall Study
Arm/Group | Pre-emptive Ethanol Lock Therapy Group | Standard Ethanol Lock Therapy Group
Started (12 infection episodes from 6 participants; 6 of these episodes (3 participants) were in both groups.) | 13; 15 Catheter Infection Episodes (Cases) (2 participants with 4 episodes of catheter infection was enrolled twice in this group.) | 14; 18 Catheter Infection Episodes (Cases) (1 participant with 2 episodes of catheter infection was enrolled twice in this group.)
Completed (Catheter Infection Episodes (Cases) reflect completed episodes with Positive blood cultures) | 4; 5 Catheter Infection Episodes (Cases) | 8; 9 Catheter Infection Episodes (Cases)
Not Completed | 9; 10 Catheter Infection Episodes (Cases) | 6; 9 Catheter Infection Episodes (Cases)
Not completed — NO POSITIVE BLOOD CULTURE | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-emptive Ethanol Lock Therapy Group | Standard Ethanol Lock Therapy Group | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 14 | 27
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay (LOS) in Those With 14 Confirmed Catheter Related Infection Cases
Description: A primary endpoint of this study is length of stay (LOS) per catheter infection episode/admission
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Population: 1 participant with 2 distinct episodes of catheter infection was enrolled twice in each group.
Measure: Mean (Standard Deviation); unit: HOURS
Units Other Than Participants: Catheter Infection Episodes (cases)
Groups:
- Pre-emptive Ethanol Lock Therapy Group: Pre-emptive Ethanol Lock Therapy Group
- Standard of Care Ethanol Lock Therapy Group: Standard of Care Ethanol Lock Therapy group
Arm/Group | Pre-emptive Ethanol Lock Therapy Group | Standard of Care Ethanol Lock Therapy Group
Number analyzed (Participants) | 4 | 8
Number analyzed (Catheter Infection Episodes (cases)) | 5 | 9
HOURS | 124 (51) | 208 (151)

2. Primary Outcome: Attributable Length of Stay (ALOS) in 14 Confirmed Catheter Related Infection Cases
Description: TIME FROM FIRST POSITIVE TO FIRST NEGATIVE BLOOD CULTURE
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Population: 1 participant with 2 distinct episodes of catheter infection was enrolled twice in each group.
Measure: Mean (Standard Deviation); unit: HOURS
Units Other Than Participants: Catheter Infection Episodes (cases)
Groups:
- Pre-emptive Ethanol Lock Therapy Group: Study Arm, given pre-emptive ELT
- Standard Ethanol Lock Therapy Group: Study Arm, given standard of care
Arm/Group | Pre-emptive Ethanol Lock Therapy Group | Standard Ethanol Lock Therapy Group
Number analyzed (Participants) | 4 | 8
Number analyzed (Catheter Infection Episodes (cases)) | 5 | 9
HOURS | 21 (20) | 32 (12)

3. Primary Outcome: Hospital COSTS in 14 Confirmed Catheter Related Infection Cases
Description: Hospital COSTS
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Population: 1 participant with 2 distinct episodes of catheter infection was enrolled twice in each group.
Measure: Mean (Standard Deviation); unit: USD $
Units Other Than Participants: Catheters
Arm/Group | Pre-emptive Ethanol Lock Therapy Group | Standard Ethanol Lock Therapy Group
Number analyzed (Participants) | 4 | 8
Number analyzed (Catheters) | 5 | 9
USD $ | 11,441 (3722) | 18,071 (3739)

4. Secondary Outcome: Catheter Sterilization
Description: Number of Catheters sterilized with interventions
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Population: 1 participant with 2 distinct episodes of catheter infection was enrolled twice in each group.
Measure: Number; unit: Catheters
Units Other Than Participants: Catheters
Arm/Group | Pre-emptive Ethanol Lock Therapy Group | Standard Ethanol Lock Therapy Group
Number analyzed (Participants) | 4 | 8
Number analyzed (Catheters) | 5 | 9
Catheters | 5 | 9

5. Secondary Outcome: Catheter Salvage
Description: Number of Infected catheters (which achieved sterilization) with salvage for at least 14 days.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Population: 1 participant with 2 distinct episodes of catheter infection was enrolled twice in each group.
Measure: Number; unit: Catheters
Units Other Than Participants: Catheters
Arm/Group | Pre-emptive Ethanol Lock Therapy Group | Standard Ethanol Lock Therapy Group
Number analyzed (Participants) | 4 | 8
Number analyzed (Catheters) | 5 | 9
Catheters | 5 | 9

6. Secondary Outcome: Number of Adverse Events Per Episode of Catheter Infection
Description: Number of Adverse events per episode of distinct catheter infection that are thought to be related to the actual study intervention, namely timing of ethanol lock placement, will be reviewed and reported for each individual infection episode/admission.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 2 weeks but up to 1 month post the last ethanol dose administration
Population: 1 participant with 2 distinct episodes of catheter infection was enrolled twice in each group.
Measure: Number; unit: Adverse Events
Units Other Than Participants: Catheter Infection Episodes (cases)
Arm/Group | Pre-emptive Ethanol Lock Therapy Group | Standard Ethanol Lock Therapy Group
Number analyzed (Participants) | 4 | 8
Number analyzed (Catheter Infection Episodes (cases)) | 5 | 9
Adverse Events | 0 | 0

7. Secondary Outcome: Re-infection
Description: Number of Re-Infected of salvaged catheters with same or new organism(s) within 28 days of prior CRI/ELT
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 2 weeks but for up to 1 month total
Population: 1 participant with 2 distinct episodes of catheter infection was enrolled twice in each group.
Measure: Number; unit: Catheters
Units Other Than Participants: Catheters
Arm/Group | Pre-emptive Ethanol Lock Therapy Group | Standard Ethanol Lock Therapy Group
Number analyzed (Participants) | 4 | 8
Number analyzed (Catheters) | 5 | 9
Catheters | 0 | 0

ADVERSE EVENTS:
Time Frame: Each participant was assessed for Adverse Events for up to 30 days post ELT receipt. (1 participant with 2 distinct episodes of catheter infection was enrolled twice in each group.)
Description: Elevation of ALT, AST from baseline; CVC line breakage, malfuntion, or thrombosis; Reinfection of line within 14 days after line.
Groups:
- Arm 1: Study Arm, given pre-emptive ELT
- Arm 2: Study Arm, given standard of care
Arm/Group | Arm 1 | Arm 2
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 0/4 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No